CLINICAL TRIAL: NCT00342303
Title: Essential Fatty Acid Metabolism in the Newborn: Equivalence of Precusors and Mediators in the Synthesis of Long Chain Polyunsaturated Fatty Acids of the n-6 and n-3 Series
Brief Title: Activity of Essential Fatty Acid Elongation/Desaturation Pathway During Early Life in Human Infants, In Vivo
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999993027; OH93-AA-N027
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-13

CONDITIONS: Fatty Acid Metabolism
Keywords: Premature Infants; Fatty Acid Metabolism; Polyunsaturated Fatty Acids; Infant Formula; Gas-chromatography; Mass Spectrometry
MeSH Terms: conditions — Premature Birth

SUMMARY:
We will test the following hypotheses:

1. The activity of the desaturating/elongating enzymes assessed by the in vivo conversion of deuterated a-linolenic and linoleic acids to DHA and AA, respectively, will be related to the duration of gestation and to postnatal age.
2. Dietary w-3 and w-6 LCPUFAs in human milk or DHA and AA supplemented formula will inhibit the desaturation/elongation of deuterated a-linolenic and linoleic acids demonstrating in vivo inhibition of the metabolic pathway by respective products.

Present evidence suggests that the parent essential fatty acids (EFA), linoleic acid (18:2 w-6) and a-linolenic acids (18:3 w-3) are insufficient to fully satisfy EFA nutrition during early life in the human. A possible need for long chain (LC, longer than 18 C chain length) EFAs in the human is suggested by the accretion rates of elongated and desaturated products in the developing fetus; the altered plasma and red cell fatty acid patterns, and the abnormal visual function observed in infants receiving solely the parent EFAs; and by the relatively high concentration of LC EFAs in human milk. Most milk formula, as compared to human milk, are lower in oleic acid, higher in linoleic, have little a-linolenic acid and virtually no LC w-3 or w-6 polyunsaturated FA (LC PUFA). This study will evaluate the capacity of human infants to form w-3 and w-6 LCPUFAs from the parent EFAs as affected by developmental stage and dietary EFA supply. The precursors will be labeled with deuterium and the products analyzed by gas chromatography / mass spectrometry GC/MS. The main products of the desaturation / elongation pathway are docosahexaenoic (DHA) and arachidonic (AA) acids for the w-3 and w-6 series, respectively. Infants will be fed human milk or formulas with or without supplemental LCPUFAs as part of a study to evaluate the effect of EFAs on CNS functional development. Infants included in this study of the effect of developmental stage on EFA desaturation/elongation will be 2-5 days of age (before any fat is administered enterally or parenterally) and 28, 32, 36 or 40 weeks gestation. In addition, infants born at 28 and 40 weeks gestation will be studied 2 and 6 weeks postnatally after dietary fat has been provided for at least 7 days and energy intake is sufficient to assure growth. To evaluate the effect of dietary EFA on DHA and AA formation we will assess elongation/ desaturation in infants receiving 3 diets: human milk (which contains w-3 and w-6 LCPUFAs); cow milk based formula providing 18:2 w-6 and 18:3 w-3 but no LCPUFAs; or formula supplemented with added LCPUFAs (DHA and AA). This study should provide new information on the effects of developmental stage and w-3 and w-6 LCPUFA supply in determining the activity of EFA elongation/desaturation in the human. This knowledge may help in improving early neonatal nutritional practices to assure meeting the EFA needs of the developing CNS.

DETAILED DESCRIPTION:
We will test the following hypotheses:

1. The activity of the desaturating/elongating enzymes assessed by the in vivo conversion of deuterated a-linolenic and linoleic acids to DHA and AA, respectively, will be related to the duration of gestation and to postnatal age.
2. Dietary w-3 and w-6 LCPUFAs in human milk or DHA and AA supplemented formula will inhibit the desaturation/elongation of deuterated a-linolenic and linoleic acids demonstrating in vivo inhibition of the metabolic pathway by respective products.

Present evidence suggests that the parent essential fatty acids (EFA), linoleic acid (18:2 w-6) and a-linolenic acids (18:3 w-3) are insufficient to fully satisfy EFA nutrition during early life in the human. A possible need for long chain (LC, longer than 18 C chain length) EFAs in the human is suggested by the accretion rates of elongated and desaturated products in the developing fetus; the altered plasma and red cell fatty acid patterns, and the abnormal visual function observed in infants receiving solely the parent EFAs; and by the relatively high concentration of LC EFAs in human milk. Most milk formula, as compared to human milk, are lower in oleic acid, higher in linoleic, have little a-linolenic acid and virtually no LC w-3 or w-6 polyunsaturated FA (LC PUFA). This study will evaluate the capacity of human infants to form w-3 and w-6 LCPUFAs from the parent EFAs as affected by developmental stage and dietary EFA supply. The precursors will be labeled with deuterium and the products analyzed by gas chromatography / mass spectrometry GC/MS. The main products of the desaturation / elongation pathway are docosahexaenoic (DHA) and arachidonic (AA) acids for the w-3 and w-6 series, respectively. Infants will be fed human milk or formulas with or without supplemental LCPUFAs as part of a study to evaluate the effect of EFAs on CNS functional development. Infants included in this study of the effect of developmental stage on EFA desaturation/elongation will be 2-5 days of age (before any fat is administered enterally or parenterally) and 28, 32, 36 or 40 weeks gestation. In addition, infants born at 28 and 40 weeks gestation will be studied 2 and 6 weeks postnatally after dietary fat has been provided for at least 7 days and energy intake is sufficient to assure growth. To evaluate the effect of dietary EFA on DHA and AA formation we will assess elongation/ desaturation in infants receiving 3 diets: human milk (which contains w-3 and w-6 LCPUFAs); cow milk based formula providing 18:2 w-6 and 18:3 w-3 but no LCPUFAs; or formula supplemented with added LCPUFAs (DHA and AA). Also, the relative efficiency of conversion of the 18-C precursors will be compared to the 20-C precursors with respect to their metabolic endpoints. This study should provide new information on the effects of developmental stage and w-3 and w-6 LCPUFA supply in determining the activity of EFA elongation/desaturation in the human. This knowledge may help in improving early neonatal nutritional practices to assure meeting the EFA needs of the developing CNS.

ELIGIBILITY:
* INCLUSION CRITERIA:

Newborns with birth weights appropriate for their gestational age born at 28, 32, 36 and 40 weeks gestation that are recovering from common neonatal morbidity will be recruited to enter the study before 5 days of age. This disease condition will not be life threatening at the time of study.

The typical disease conditions expected based on the pilot phase of study are infants recovering from asphyxia, infants recovering from transient tachypnea, infants recovering from suspect pneumonia, infants recovering from hyaline membrane disease.

Hyperbilirubinemia in conjunction with disease condition will not be a reason for exclusion.

Newborns with birth weights below the tenth percentile of the weight distribution for a given gestational age born at 30-34 and 36-38 weeks gestation.

Will include infants born at 28 to 40 weeks who are free of major neonatal morbidity and will be recruited to enter the study at 10 days of age.

EXCLUSION CRITERIA:

Maternal factors which may affect their fatty acid metabolism of the neonate.

* Vegetarian or vegan diet during pregnancy
* Metabolic disease which may affect essential fatty acid status of the fetus (hyperlipidemia, diabetes)

Postnatal factors:

Birth weight inadequate for gestational age (birth weight below the 10th percentile or above the 90th percentile for gestational age)

Significant acute neonatal morbidity which interferes with normal lipid metabolism during the study period. Infants who are recovering from common neonatal morbidities that do not have obvious effects on elongase/desaturase activity will not be excluded.

Feeding other than prescribed for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 1993-06-08; Study Completion 2010-07-13

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Clinica Presbiteriana Madre Hijo, Santiago
  - Hospital Luis Tisne, Santiago

REFERENCES:
- [Background] Lee AG, East JM, Froud RJ. Are essential fatty acids essential for membrane function? Prog Lipid Res. 1986;25(1-4):41-6. doi: 10.1016/0163-7827(86)90009-3. No abstract available. PMID 2962202
- [Background] Glomset JA. Fish, fatty acids, and human health. N Engl J Med. 1985 May 9;312(19):1253-4. doi: 10.1056/NEJM198505093121909. No abstract available. PMID 3990716
- [Background] Sprecher H. Biochemistry of essential fatty acids. Prog Lipid Res. 1981;20:13-22. doi: 10.1016/0163-7827(81)90009-6. No abstract available. PMID 7342077